CLINICAL TRIAL: NCT03839238
Title: Safety Observation on Human Embryonic Stem Cell (hESC) Derived Mesenchymal Stem Cells(MSC) Like Cell for the Meniscus Injury
Brief Title: Safety Observation on hESC Derived MSC Like Cell for the Meniscus Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wuhan Tongji Hospital
Record Dates: First submitted 2018-11-28; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-11

CONDITIONS: Meniscus Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meniscus Injured patients (Experimental): hESC Derived MSC Like Cell
  Interventions: Biological: hESC derived MSC like cell

INTERVENTIONS:
Biological: hESC derived MSC like cell — Different dosage of hESC derived MSC like cell for the meniscus injured patients

SUMMARY:
human embryonic stem cell derived mesenchymal stem cells like cell for the meniscus injury, and observe the safety of the cells for meniscus injury

DETAILED DESCRIPTION:
Three different dosage of human embryonic stem cell derived mesenchymal stem cells like for meniscus injury patients, and observe the safety of the cells for meniscus injury.

ELIGIBILITY:
Inclusion Criteria:

* Grade Ⅰ-Ⅱ meniscus injury of knee joint
* The patients who still have the pain of knee joint and/or limitation of the function after accepted 3 months of nonoperative treatment

Exclusion Criteria:

* Recent history of lower limb fractures or intra-articular drug injection
* The patients who have meniscus injury of knee joint need the surgical repair
* The patients who have the severe coagulation disorders, cardiopulmonary failure and so on
* The women who are pregnant or nursing
* There are electronic implants such as pacemakers in the body
* The patients who are infected the HIV, the virus of hepatitis or syphilis
* The patients who are alcoholism or drug user
* The patients who have vestibular and balance disorders
* The patients with severe cognitive impairment who cannot follow instructions to complete the treatment
* The patients who don't sign the informed consent
* The patients who have tumor
* Immunodeficiency patients
* The patients who have congenital or acquired knee malformation
* Patients or researchers who are participating in other clinical trials believe that other reasons are not appropriate for clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in number of adverse events based on the National Cancer Institute-Common Terminology Criteria for Adverse Events | 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  Adverse events include：allergic reactions, local reactions or infections at the injection site and muscle or skeletal dysplasia

SECONDARY OUTCOMES:
Ultrasound of knee joint | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  Ultrasound of knee joint
Visual Analog Score for pain（VAS） | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  VAS is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective pain. The scale range is from 0 to 10, the higher the score, the more severe the pain.
Range of knee motion | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  to use the goniometer to measure the range of knee motion
Lysholm Knee Scale | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  The scale is to assess the function of knee. The scale range is from 0 to 100, the higher the score, the more severe the knee problems. This scale includes 8 items, and the total score is the sum of these 8 items' scores. Individual items are scored differently, using individual scoring scales: 1. limp (0,3,5), 2. support (0,2,5), 3. locking (0,2,6,10,15), 4. instability (0,5,10,15,20,25), 5. pain (0,5,10,15,20,25), 6. swelling (0,2,6,10), 7. stair climbing (0,2,6,10), 8. squatting (0,2,4,5).
MRI of knee | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  MRI of knee
Global posture analysis system | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  to test the static balance
Dynamic balance test | baseline, 1 week, 1 month, 2months and 3 months after the injection of MSC Like Cell
  Use the dynamic posture evaluator

CONTACTS AND LOCATIONS:
Overall Officials: Hong Chen, Doctor, Study Director — Wuhan TongJi Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College of Science and Technology, Wuhan, Hubei, China